CLINICAL TRIAL: NCT02556853
Title: Comparison Between Ultrasound and Clinical Assessment of the Correct Positioning of Left Double Lumen Endotracheal Tube
Brief Title: Ultrasound for Double Lumen Endotracheal Tube
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Thoracic Surgery Department has almost stopped completely its surgical activities and the completion of the study doesn't seem to be feasible.
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Georgios Kotsovolis, Doctor, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14074
Record Dates: First submitted 2015-09-20; First posted 2015-09-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lung Ultrasound
Keywords: Ultrasound; Double lumen tube

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Determination of correct placement of the double lumen tube by lung ultrasound.
  Interventions: Device: Determination of tube position by ultrasound.
- Clinical (Active Comparator): Determination of correct placement of the double lumen tube by clinical examination.
  Interventions: Other: Determination of tube position by auscultation.

INTERVENTIONS:
Device: Determination of tube position by ultrasound. — After placement of the left sided double lumen endotracheal tube, ventilation of both lungs will be verified by ultrasound (Sonoscape S6®). The ultrasound probe will be placed between the 2nd and 3rd intercostal space at the level of the midclavicular line parallel to the line. The probe will be slightly moved or tilted until the pleural line is identified. If lung sliding is identified then the ventilation of the lung will be considered adequate. The same procedure will be repeated for each lung alone, after lung separation is applied. Verification of the ultrasound findings will be performed by bronchoscopy (Pentax®). The depth of the tube will be adjusted according to the bronchoscopy findings until correct positioning is established.
  Arms: Ultrasound
Other: Determination of tube position by auscultation. — After placement of the left sided double lumen endotracheal tube, ventilation of both lungs will be verified by auscultation of the upper lung fields. The same procedure will be repeated for each lung alone, after lung separation is applied. Verification of the ultrasound findings will be performed by bronchoscopy (Pentax®). The depth of the tube will be adjusted according to the bronchoscopy findings until correct positioning is established.
  Arms: Clinical

SUMMARY:
The patients will be allocated to 2 groups: the ultrasound group and the clinical group. The correct position of the double lumen tube will be determined by ultrasound (Sonoscape S6®) for the patients of the one group (group U) and by clinical examination for the patients of the other group (group C). The correct placement will be verified by bronchoscopy (Pentax®). The two methods will be compared in terms of sensitivity and specificity. The main purpose of the study is to determine if the ultrasound can be used for determination of the correct placement of the left sided double lumen endotracheal tube

ELIGIBILITY:
Inclusion Criteria:

* Surgery requiring placement of double-lumen endotracheal tube.
* ASA 1-3

Exclusion Criteria:

* History of difficult or impossible intubation.
* Clinical findings of possible difficult intubation according to the standard preoperative airway assessment.
* Impossible placement of a double lumen tube

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Correct position of the tube (yes/no). | Within an average of 5 minutes after the placement of the double lumen tube
  The anesthesiologist who will place the left-sided double lumen tube will determine if the position of the tube is correct according to the ultrasound or clinical findings.
Correct position of the tube by bronchoscopy (yes/no). | Within an average of 10 minutes after the placement of the double lumen tube.
  After the assessment of the tube's position, a second anesthesiologist will verify the position of the tube by bronchoscopy.

SECONDARY OUTCOMES:
Time needed | Within an average of 10 minutes after the placement of the double lumen tube.
  The total time passed from the beginning of laryngoscopy until the final verification of the tube's position.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia department; 424 Army General Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Sustic A, Protic A, Cicvaric T, Zupan Z. The addition of a brief ultrasound examination to clinical assessment increases the ability to confirm placement of double-lumen endotracheal tubes. J Clin Anesth. 2010 Jun;22(4):246-9. doi: 10.1016/j.jclinane.2009.07.010. PMID 20522353
- [Background] Sustic A, Miletic D, Protic A, Ivancic A, Cicvaric T. Can ultrasound be useful for predicting the size of a left double-lumen bronchial tube? Tracheal width as measured by ultrasonography versus computed tomography. J Clin Anesth. 2008 Jun;20(4):247-52. doi: 10.1016/j.jclinane.2007.11.002. PMID 18617120
- [Background] Alvarez-Diaz N, Amador-Garcia I, Fuentes-Hernandez M, Dorta-Guerra R. Comparison between transthoracic lung ultrasound and a clinical method in confirming the position of double-lumen tube in thoracic anaesthesia. A pilot study. Rev Esp Anestesiol Reanim. 2015 Jun-Jul;62(6):305-12. doi: 10.1016/j.redar.2014.06.005. Epub 2014 Aug 20. English, Spanish. PMID 25149114